CLINICAL TRIAL: NCT01738087
Title: A Phase II, Monocentric, Open, Randomized, 6-way Cross-over Clinical Pharmacology Study to Evaluate the Lung Bioavailability of BDP/B17MP and Formoterol and the Total Systemic Exposure Across Two Different Strengths of CHF 1535 NEXThaler Dry Powder Inhaler (Fixed Combination of Beclomethasone Dipropionate Plus Formoterol Fumarate 100/6 mcg and 200 mcg) Administered With and Without Activated Charcoal in Adult Asthmatic Patients.
Brief Title: Lung Bioavailability and Total Systemic Exposure to Beclomethasone17MonoPropionate and Formoterol Across Two Strengths of NEXThaler Inhalation Powder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-1205-PR-0087; 2012-002370-30 (EudraCT Number)
Record Dates: First submitted 2012-11-15; First posted 2012-11-30 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Asthmatic
Keywords: patients; Adult
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- NEXThaler 100/6 mcg DPI (Experimental): Single dose (4 inhalations)of NEXThaler 100/6 mcg DPI: total dose 400/24 mcg
  Interventions: Drug: NEXThaler 100/6 mcg DPI
- NEXThaler 200/6 mcg DPI (Experimental): Single dose (4 inhalations)of NEXThaler 200/6 mcg DPI: total dose: 800/24 mcg
  Interventions: Drug: NEXThaler 200/6 mcg DPI
- NEXThaler placebo (Placebo Comparator): Single dose (4 inhalations)
  Interventions: Drug: NEXThaler placebo
- NEXThaler 100/6 mcg plus CB (Experimental): Single dose (4 inhalations) NEXThaler 100/6 mcg administered with activated charcoal (Charcoal Block): total dose 400/24 mcg
  Interventions: Drug: NEXThaler 100/6 mcg DPI
- NEXThaler 200/6 mcg plus CB (Experimental): Single dose (4 inhalations) NEXThaler 200/6 mcg administered with activated charcoal (Charcoal Block): total dose 800/24 mcg
  Interventions: Drug: NEXThaler 200/6 mcg DPI
- Flixotide Accuhaler 500 mcg (Active Comparator): Single dose (2 inhalations) of fluticasone propionate
  Interventions: Drug: Flixotide Accuhaler 500 mcg

INTERVENTIONS:
Drug: NEXThaler 100/6 mcg DPI
  Other Names: Fixed combination of BDP plus formoterol fumarate
  Arms: NEXThaler 100/6 mcg DPI; NEXThaler 100/6 mcg plus CB
Drug: Flixotide Accuhaler 500 mcg — Active comparator
  Other Names: Fluticasone Propionate
  Arms: Flixotide Accuhaler 500 mcg
Drug: NEXThaler 200/6 mcg DPI
  Other Names: Fixed combination of BDP plus formoterol fumarate
  Arms: NEXThaler 200/6 mcg DPI; NEXThaler 200/6 mcg plus CB
Drug: NEXThaler placebo — Placebo comparator
  Arms: NEXThaler placebo

SUMMARY:
The study is aimed to assess the dose proportional total systemic exposure (when the administration is without the activated charcoal) to B17MP (active metabolite of BDP) and its lung bioavailability (when the administration is with the activated charcoal) after single inhalation of CHF 1535 NEXThaler DPI at two dose strengths.

At the same time, the study will assess if the lung deposition and the total systemic exposure to Formoterol is affected by increasing doses of BDP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma as defined by Global Initiative for Asthma (GINA) 2011
* Asthmatic patients already treated with low daily doses of Inhaled Corticosteroids (ICS) (eg budesonide or equivalent lower than 400 mcg/day) or low dose of ICS/Long Acting Beta2 Agonists (LABA) fixed combinations.
* Patients with Forced Expiratory Volume in 1 sec (FEV1) >= 70 % of predicted values
* Non or ex-smokers
* Body Mass Index (BMI) >= 18.5 and <= 32 kg/m2

Exclusion Criteria:

* Pregnant or lactating women unless using acceptable methods of contraception
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* History of near fatal asthma
* Patients with abnormal QTcF at screening Visit
* Hospitalization due to asthma exacerbation within 4 weeks prior to the screening visit or during the run-in period.
* Lower respiratory tract infection within 4 weeks prior to the screening visit or during the run-in period.
* History of drug addiction or excessive use of alcohol ;
* Diagnosis of restrictive lung disease.
* Patients treated with oral or parenteral corticosteroids in the previous 2 months before the screening visit (3 months for parenteral depot corticosteroids)
* Significant medical history or any laboratory abnormality indicative of a significant underlying condition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Formoterol AUC0-t and B17MP AUC0-t | from predose until 12 hr post dose

SECONDARY OUTCOMES:
BDP pharmacokinetic (PK) parameters | from predose until 12 hr post dose
  The following parameters will be evaluated: AUC0-t, AUC0-12h, AUC0-inf, Cmax, tmax, t1/2
Other PK parameter of B17MP and formoterol | from predose until 12 hours postdose
  the following pharmacokinetic parameters will be evaluated: AUC0-12, AUCinf, Cmax, tmax, t1/2

OTHER OUTCOMES:
Plasma glucose | from predose until 12 hours postdose
  the following parameters will be evaluated: AUC0-4h, AUC0-12h, Cmax and tmax
Heart rate (HR) | from predose until 12 hours postdose
  the following parameters will be evaluated: HR AUC0-12/12h
Plasma cortisol | from predose until 24 hours postdose
  the following parameters will be evaluated: AUC0-24, Cmin and tmin
Plasma potassium | from predose until 12 hours postdose
  the following parameters will be evaluated: AUC0-4h, AUC0-12h, Cmin ad tmin
Systolic and Diastolic Blood Pressure (SBP and DBP) | from predose until 12 hours postdose
  the following parameters will be evaluated: SBP AUC0-12/12h and DBP AUC0-12/12h

CONTACTS AND LOCATIONS:
Locations (1):
- The Medicine Evaluation Unit, Manchester, United Kingdom

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2012-002370-30
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-1205-PR-0087.pdf